CLINICAL TRIAL: NCT03811847
Title: A Pilot, Multiple Crossover, Randomized Block Sequence, Double-Blind, Placebo-Controlled Trial for Use of Methylphenidate for Cognitive and Behavioral Symptoms in Mild Cognitive Impairment and Dementia
Brief Title: A Pilot of Methylphenidate in Mild Cognitive Impairment and Dementia Participants.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven E Arnold, MD, Managing Director Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2018P003099
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Dementia
MeSH Terms: conditions — Alzheimer Disease | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: The study uses a double-blinded, multi-crossover, randomized controlled trial design. This type of trial design in AD allow for each subject to serve as their own control as they progress through several randomized blocks of experimental treatment and placebo. Thus, multi-crossover studies carried out with systemically applied outcome measures, pre-specified doses of study drug, and washout periods serve as unbiased estimates of treatment effect for individual subjects. When data from several subjects are analyzed together following such a N-of-1 design, substantial increases in statistical power is afforded with a fraction of the subjects and assessments required for similar levels of power in conventional parallel group trials. There are 6 different block randomization sequences for which subjects were assigned.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH (Experimental): Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received Methylphenidate (MPH) for 2 weeks, then placebo for 2 weeks, then MPH for 2 weeks, then Placebo for 2 weeks, then Placebo for 2 weeks, then MPH for 2 weeks.
  Interventions: Drug: Methylphenidate Extended Release Oral Capsule; Other: Placebo
- Sequence 2:MPH, PBO, PBO, MPH, MPH, PBO (Experimental): Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received Methylphenidate (MPH) for 2 weeks, then placebo for 2 weeks, then PBO for 2 weeks, then MPH for 2 weeks, then MPH for 2 weeks, then PBO for 2 weeks.
  Interventions: Drug: Methylphenidate Extended Release Oral Capsule; Other: Placebo
- Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH (Experimental): Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received Methylphenidate (MPH) for 2 weeks, then placebo for 2 weeks, then MPH for 2 weeks, then Placebo for 2 weeks, then Placebo for 2 weeks, then MPH for 2 weeks.
  Interventions: Drug: Methylphenidate Extended Release Oral Capsule; Other: Placebo
- Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO (Experimental): Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received PBO for 2 weeks, then MPH for 2 weeks, then MPH for 2 weeks, then Placebo for 2 weeks, then MPH for 2 weeks, then PBO for 2 weeks.
  Interventions: Drug: Methylphenidate Extended Release Oral Capsule; Other: Placebo
- Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH (Experimental): Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received PBO for 2 weeks, then MPH for 2 weeks, then MPH for 2 weeks, then Placebo for 2 weeks, then Placebo for 2 weeks, then MPH for 2 weeks.
  Interventions: Drug: Methylphenidate Extended Release Oral Capsule; Other: Placebo
- Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO (Experimental): Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received PBO for 2 weeks, then MPH for 2 weeks, then PBO for 2 weeks, then MPH for 2 weeks, then MPH for 2 weeks, then PBO for 2 weeks.
  Interventions: Drug: Methylphenidate Extended Release Oral Capsule; Other: Placebo

INTERVENTIONS:
Drug: Methylphenidate Extended Release Oral Capsule — Stimulant It can treat ADHD and narcolepsy.
  1 capsule 18mg
  Other Names: Ritalin
Other: Placebo — Placebo comparator MPH Matched Placebo Tablet

SUMMARY:
Investigators are doing this research study to find out if methylphenidate (MPH) can help people with Mild Cognitive Impairment (MCI) or mild dementia likely due to Alzheimer's Disease (AD) and related disorders (ADRD).

The study drug MPH is approved by the U.S. Food and Drug Administration (FDA) to treat Attention Deficit/Hyperactivity Disorder (ADHD), but MPH is not approved by the FDA to treat Mild Cognitive Impairment or mild dementia related to Alzheimer's Disease. However, other studies have been done in which MPH has been given to people with neurodegenerative dementias and results have shown some improvement in these people's mood and cognition. Investigators would like to see if MPH will help mood and cognition.

This study will take place completely virtually (with the option to come in for the first visit to meet the study team). All study visits will occur over a secure videoconferencing platform. All study materials will be shipped directly to the home of each participant.

DETAILED DESCRIPTION:
Investigators will give participants a supply of study drug. Participants will take the study drug by mouth once a day for 16 weeks. It is important for participants to follow our instructions about how to take the study drug. Participants can take the drug with or without food. Investigators will provide enough study drug for participants to take until the next visit.

For this study, there are 3 blocks: each month-long block will consist of MPH for a two-week period (I.e. "A" Blocks 1, 2, 3) and PBO for a two-week period (I.e. "B" Blocks 1, 2, 3) in random assignment order for each block. Thus, all volunteers will receive a four-week PBO-lead in and acclimatization followed by treatment with MPH or matching PBO for eight-weeks each in three randomized sequence crossover blocks for a total of 10 weeks of PBO and 6 weeks of MPH.

Weekly Tasks During the study, certain tasks must be done each week.

Every Day:

The following tasks must be done each day throughout the study:

* Wear the activity tracker
* Take study medication

Six Days per Week:

The following tasks will be completed six days per week:

* Complete online cognitive games

  o Use online brain games to rate daily mood and sleep quality
* Synchronize Fitness tracker to study provided tablet (if requested)

Once every five days:

The following activities must be done approximately every five days throughout the trial:

• Charge Fitness tracker during a time when the subject is resting but not sleeping

The study coordinator will periodically log into both the Fitness tracker dashboard and the online brain game account to check the battery level of the Fitness tracker, ensure the Fitness tracker is synching to the Fitness tracker dashboard, and monitor the completion of cognitive exercises.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects meeting all of the following criteria will be allowed to enroll in the study:

  1. Aged 55-95 inclusive;
  2. Diagnosis of MCI or mild-stage dementia presumed due to AD and AD-related disorders;
  3. Cognitive abilities sufficient to be able to complete all study tasks as determined by the PI or a Co-I;
  4. Education level, English language skills, and literacy that indicates participant will be able to comprehend all assessments;
  5. Neuropsychiatric Inventory Agitation/Aggression Question 4 = "No" or "Yes" with a mild severity rating.
  6. Willing and able to complete all assessments and study procedures;
  7. Not pregnant, lactating, or of child-bearing potential
  8. Volunteer has a Study Partner with at least two days per week of contact and willing to complete partner study forms;
  9. No exclusionary medications or dietary supplements. See Section 6.5.8.1
  10. If on cholinesterase inhibitor and/or memantine, doses are stable for 3 months prior to baseline.
  11. Basic video conferencing capabilities and a willingness to participate in a virtual trial (including self-administration of ECG).

Exclusion Criteria:

* Subjects meeting any of the following criteria during the screening evaluation will be excluded:

  1. Any history of specific CNS disease other than AD or AD-related disorders, such as major clinical stroke, brain tumor, normal pressure hydrocephalus, multiple sclerosis, significant head trauma with persistent neurological or cognitive deficits or complaints;
  2. Clinically significant or unstable medical condition that could affect safety or compliance with the study and would, in the opinion of the investigator, pose a risk to the participant if they were to participate in the study;
  3. Major active or chronic psychiatric illness (e.g. depression, bipolar disorder, obsessive compulsive disorder, schizophrenia) within the previous year;
  4. Current suicidal ideation or history of suicide attempt;
  5. History of alcohol or other substance abuse or dependence with the past two years;
  6. Clinically significant abnormalities on complete blood count, comprehensive metabolic panel, B12, or TSH screening safety lab results;
  7. Concomitant use of medications with psychoactive properties that may deleteriously affect cognition (anticholinergics, antihistamines, antipsychotics, sedative hypnotics, anxiolytics);
  8. Treatment with monoamine oxidase inhibitors, coumadin, phenobarbital, phenytoin, primidone, tricyclic antidepressants or other medicines with potential for clinically significant interaction;
  9. Hypersensitivity to MPH;
  10. History of marked anxiety and agitation, ADHD, motor tics, glaucoma, or a history or family history of Tourette's Syndrome;
  11. Clinically significant cardiac condition for which MPH may be contradicted as determined by study physician, such as MI or ventricular arrhythmia within 6 months of enrollment;
  12. History of untreated, uncontrolled hypertension or a blood pressure greater than 150/90 during the screening period;
  13. Use of other small molecule or device- based investigational agents one month prior to entry and for the duration of the trial.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Arnold, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Clinical Translational Research Unit, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DesRuisseaux LA, Williams VJ, McManus AJ, Gupta AS, Carlyle BC, Azami H, Gerber JA, Bolling AM, Cook CL, Betensky RA, Arnold SE. A pilot protocol to assess the feasibility of a virtual multiple crossover, randomized controlled trial design using methylphenidate in mild cognitive impairment. Trials. 2020 Dec 11;21(1):1016. doi: 10.1186/s13063-020-04752-x. PMID 33308285

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 Participants signed consent and enrolled. 3 Screen failed and 1 Withdrew due to study non compliance, prior to assignment to groups. 7 participants proceeded to assignment and Block 1A.
Groups:
- Experimental: Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH: Experimental: Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH
  Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received Methylphenidate (MPH) for 2 weeks, then placebo for 2 weeks, then MPH for 2 weeks, then Placebo for 2 weeks, then Placebo for 2 weeks, then MPH for 2 weeks.
- Experimental: Sequence 2:MPH, PBO, PBO, MPH, MPH, PBO: Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received Methylphenidate (MPH) for 2 weeks, then placebo for 2 weeks, then PBO for 2 weeks, then MPH for 2 weeks, then MPH for 2 weeks, then PBO for 2 weeks.
- Experimental: Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH: Experimental: Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received Methylphenidate (MPH) for 2 weeks, then placebo for 2 weeks, then MPH for 2 weeks, then Placebo for 2 weeks, then Placebo for 2 weeks, then MPH for 2 weeks.
- Experimental: Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO: Experimental: Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received PBO for 2 weeks, then MPH for 2 weeks, then MPH for 2 weeks, then Placebo for 2 weeks, then MPH for 2 weeks, then PBO for 2 weeks.
- Experimental: Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH: Experimental: Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received PBO for 2 weeks, then MPH for 2 weeks, then MPH for 2 weeks, then Placebo for 2 weeks, then Placebo for 2 weeks, then MPH for 2 weeks.
- Experimental: Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO: Experimental: Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO Over the 16-week study, each participant moved through four, 4-week treatment periods: a Placebo (PBO) lead-in, acclimation period followed by three, crossover Methylphenidate (MPH) vs PBO "blocks". Each "block" consisted of treatment with MPH for two-weeks and treatment with PBO for two-weeks; each block order will be randomly assigned. In this group, participants first received PBO for 2 weeks, then MPH for 2 weeks, then PBO for 2 weeks, then MPH for 2 weeks, then MPH for 2 weeks, then PBO for 2 weeks.
Period: Block 1A
Arm/Group | Experimental: Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH | Experimental: Sequence 2:MPH, PBO, PBO, MPH, MPH, PBO | Experimental: Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH | Experimental: Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO | Experimental: Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH | Experimental: Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO
Started | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Block 1B
Arm/Group | Experimental: Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH | Experimental: Sequence 2:MPH, PBO, PBO, MPH, MPH, PBO | Experimental: Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH | Experimental: Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO | Experimental: Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH | Experimental: Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO
Started | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Block 2 A
Arm/Group | Experimental: Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH | Experimental: Sequence 2:MPH, PBO, PBO, MPH, MPH, PBO | Experimental: Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH | Experimental: Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO | Experimental: Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH | Experimental: Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO
Started | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Block 2B
Arm/Group | Experimental: Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH | Experimental: Sequence 2:MPH, PBO, PBO, MPH, MPH, PBO | Experimental: Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH | Experimental: Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO | Experimental: Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH | Experimental: Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO
Started | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Block 3A
Arm/Group | Experimental: Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH | Experimental: Sequence 2:MPH, PBO, PBO, MPH, MPH, PBO | Experimental: Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH | Experimental: Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO | Experimental: Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH | Experimental: Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO
Started | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Block 3B
Arm/Group | Experimental: Sequence 1:MPH, PBO, MPH, PBO, PBO, MPH | Experimental: Sequence 2:MPH, PBO, PBO, MPH, MPH, PBO | Experimental: Sequence 3:MPH, PBO, PBO, MPH, PBO, MPH | Experimental: Sequence 4:PBO, MPH, MPH, PBO, MPH, PBO | Experimental: Sequence 5: PBO, MPH, MPH, PBO, PBO, MPH | Experimental: Sequence 6: PBO, MPH, PBO, MPH, MPH, PBO
Started | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were analyzed in treatment/placebo groups based on randomized crossover assignment.
Groups:
- Randomized Crossover Methylphenidate/Placebo: During this study, participants will get both the study drug Methylphenidate Extended Release Capsule and the placebo in random order. Placebo is being used in this study to compare to see if any improvements in cognition other areas are due to the study drug or due to other reasons.
  Methylphenidate Extended Release Oral Capsule: Stimulant It can treat ADHD and narcolepsy.
Arm/Group | Randomized Crossover Methylphenidate/Placebo
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.57 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of a Virtual Multicrossover Randomized Control Trial Design as Measured my Completion Rates and Medication Compliance.
Description: To assess feasibility of this study design, completion rates of all study tasks and medication dosing will be evaluated. Benchmark goals for feasibility measures are set as follows: retain >80% of participants enrolled, observe >80% medication adherence, and >80% outcome assessment completion rates.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: During this study, participants will get both the study drug Methylphenidate Extended Release Capsule and the placebo in random order.
  For this study, there are 3 blocks: each month-long block will consist of MPH for a two-week period (I.e. Blocks 1a, 2a, 3a) and PBO for a two-week period (I.e. Blocks 1b, 2b, 3b) in random assignment order for each block. Thus, all volunteers will receive a four-week PBO-lead in and acclimatization followed by treatment with MPH or matching PBO for eight-weeks each in three randomized sequence crossover blocks for a total of 10 weeks of PBO and 6 weeks of MPH.
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Participants
  Participant retention | 7
  Medication Compliance | 7
  Assessment completion | 7

2. Secondary Outcome: Cognition as Measured by the Repeatable Battery for the Assessment Neuropsychological Status-Update (RBANS)
Description: This study is investigating the effects of methylphenidate to see if it will help improve cognition in adults with Alzheimer's Disease. RBANS scores range from 40 to 160 with higher scores indicating higher cognitive functioning.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: scores on scale
Groups:
- Study Participants on MPH Treatment: Study Participants on MPH Treatment Blocks
- Study Participants on PBO Block: Study Participants on Placebo Blocks
Arm/Group | Study Participants on MPH Treatment | Study Participants on PBO Block
Number analyzed (Participants) | 7 | 7
scores on scale | 68.8 (14.1) | 70.7 (13.0)

3. Secondary Outcome: Cognition as Measured by Daily, Home-based Brain Games (Lumosity, Lumos Labs, Inc.)
Description: This study is investigating the effects of methylphenidate to see if it will help improve cognition in adults with Alzheimer's Disease using daily Lumosity brain games. The range of possible Lumosity scores varies, but higher scores indicate better game performance. LPI (Lumosity Performance Index) is a standardized performance metric that shows how well you are performing on Lumosity games and lets you compare performance across games and Cognitive Areas. Cognitive LPI is calculated using a weighted average of the Game LPIs from all Cognitive Areas. LPI: The low score is 0, the high score is 2000. Average is 1000.
Time Frame: 4 months
Population: 6 participants played Lumosity games. LPI values for all 12 games were averaged into an LPI Composite Score for each participant in each treatment phase (MPH or PBO) in each block (1,2,3), then averaged the LPI composites for each treatment condition (MPH or PBO) for each individual, and then averaged the individuals for each treatment condition and got the standard deviation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Study Participants on MPH Blocks: Study Participants on MPH Treatment Blocks
- Study Participants on Placebo: Study Participants on PBO Blocks
Arm/Group | Study Participants on MPH Blocks | Study Participants on Placebo
Number analyzed (Participants) | 6 | 6
scores on a scale | 465.8 (308.4) | 451.6 (291.1)

4. Secondary Outcome: Sleep as Measured by Fitbit Charge 3
Description: This study is investigating whether treatment with methylphenidate affects sleep levels. Methylphenidate may increase daily activity or affect the amount or quality of sleep.
Time Frame: 4 months
Population: Data was not collected.
Groups:
- Participants on MPH Block: Fit bit Data from participants while on Methylphenidate treatment block
- Participants on PBO Block: Fit bit Data from participants while on PBO treatment block
Arm/Group | Participants on MPH Block | Participants on PBO Block
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Activity Level as Measured by Fitbit During MPH/PBO Blocks
Description: Activity level as measured by the fitbit during MPH/Placebo blocks
Time Frame: 4 months
Population: Data was not collected.
Groups:
- Activity While Participants on MPH Treatment Block: Fit bit Data from participants while on Methylphenidate treatment block
- Activity While Participants on Placebo Block: Fit bit Data from participants while on PBO treatment block
Arm/Group | Activity While Participants on MPH Treatment Block | Activity While Participants on Placebo Block
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from each participant up to 18 weeks
Groups:
- AEs While Participants on MPH Treatment Block: AEs that occurred while participants were on Methylphenidate treatment block
- AEs While Participants on Placebo Block: AEs that occurred while participants were on Placebo block
Arm/Group | AEs While Participants on MPH Treatment Block | AEs While Participants on Placebo Block
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEs While Participants on MPH Treatment Block (N=7) | AEs While Participants on Placebo Block (N=7)
insomnia (Nervous system disorders) | 2 (4) | 2 (4)
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
anxiety (Nervous system disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03811847/Prot_SAP_000.pdf